CLINICAL TRIAL: NCT01594749
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Parallel-Group Study, Conducted Under In-House Blinding Conditions, to Examine the Efficacy and Safety of a Single 150 mg Dose of Intravenous Fosaprepitant Dimeglumine for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) Associated With Moderately Emetogenic Chemotherapy
Brief Title: Efficacy and Safety of Fosaprepitant Dimeglumine in Preventing Chemotherapy-Induced Nausea and Vomiting (MK-0517-031)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0517-031
Record Dates: First submitted 2012-04-24; First posted 2012-05-09 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV)
Keywords: NK-1 Receptor Antagonist, CINV, Emesis, MEC
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant; Aprepitant; Dexamethasone; Calcium Dobesilate; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosaprepitant Regimen (Experimental): On Day 1, participants received fosaprepitant, 150 mg intravenous (IV) infusion, ~30 minutes prior to chemotherapy PLUS dexamethasone 12 mg, orally (PO) ~30 minutes prior to chemotherapy PLUS ondansetron 16 mg total dose: 8 mg PO ~30-60 minutes prior to chemotherapy, followed by 8 mg PO, 8 hours after first dose PLUS dexamethasone placebo, PO ~30 minutes prior to chemotherapy. On Days 2 and 3, participants received ondansetron placebo, PO every 12 hours. Rescue Therapy: For established cases of nausea or vomiting, medications may have been prescribed from these permitted choices: 5-HT3 antagonists (granisetron, dolasetron, tropisetron or ondansetron); phenothiazines (e.g. prochlorperazine, fluphenazine, perphenazine, thiethylperazine, or chlorpromazine); butyrophenones (e.g. haloperidol or droperidol); benzamides (e.g. metoclopramide or alizapride); benzodiazepines; corticosteroids; domperidone.
  Interventions: Drug: Fosaprepitant dimeglumine; Drug: Dexamethasone; Drug: Ondansetron; Drug: Dexamethasone Placebo; Drug: Ondansetron Placebo; Drug: Rescue Therapy
- Control Regimen (Active Comparator): On Day 1, participants received fosaprepitant placebo, 150 mL IV infusion, ~30 minutes prior to chemotherapy PLUS dexamethasone 20 mg, PO ~30 minutes prior to chemotherapy PLUS ondansetron 16 mg total dose: 8 mg PO ~30-60 minutes prior to chemotherapy; followed by 8 mg PO, 8 hours after the first dose. On Days 2-3, participants received ondansetron 8 mg, PO every 12 hours. Rescue Therapy: For established cases of nausea or vomiting, medications may have been prescribed from these permitted choices: 5-HT3 antagonists (granisetron, dolasetron, tropisetron or ondansetron); phenothiazines (e.g. prochlorperazine, fluphenazine, perphenazine, thiethylperazine, or chlorpromazine); butyrophenones (e.g. haloperidol or droperidol); benzamides (e.g. metoclopramide or alizapride); benzodiazepines; corticosteroids; domperidone.
  Interventions: Drug: Fosaprepitant Placebo; Drug: Dexamethasone; Drug: Ondansetron; Drug: Rescue Therapy

INTERVENTIONS:
Drug: Fosaprepitant dimeglumine
  Other Names: EMEND for Injection; MK-0517
  Arms: Fosaprepitant Regimen
Drug: Fosaprepitant Placebo
  Arms: Control Regimen
Drug: Dexamethasone
  Other Names: Decadron
Drug: Ondansetron
  Other Names: Zofran
Drug: Dexamethasone Placebo
  Arms: Fosaprepitant Regimen
Drug: Ondansetron Placebo
  Arms: Fosaprepitant Regimen
Drug: Rescue Therapy

SUMMARY:
This study aims to demonstrate that, when given concomitantly with a 5-hydroxytryptamine 3 (5-HT3) antagonist and a corticosteroid, a single 150 mg intravenous (IV) dose of fosaprepitant given on Day 1 is superior to the control regimen of 5-HT3 antagonist and corticosteroid only, in preventing chemotherapy-induced nausea and vomiting (CINV) associated with moderately emetogenic chemotherapy (MEC).

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed malignant disease
* Is naive to moderately and highly emetogenic chemotherapy
* Is scheduled to receive a single IV dose of one or more MEC agents on Day 1, except for the combination of anthracycline and cyclophosphamide
* Has a predicted life expectancy of at least 4 months, and a Karnofsky score of at least 60 indicating that the participant requires occasional assistance, but is able to care for most of his/her needs.
* Female of childbearing potential demonstrates a negative urine pregnancy test, and agrees to remain abstinent or use two acceptable forms of birth control for at least 14 days prior to study, throughout the study, and at least 1 month following last dose of study drug.

Exclusion Criteria:

* Has vomited in the 24 hours prior to treatment Day 1
* Has symptomatic primary or metastatic symptomatic central nervous system malignancy causing nausea and/or vomiting
* Is scheduled to receive chemotherapy agent classified as highly emetogenic
* Has received or will receive total body irradiation, or radiation therapy to the abdomen, pelvis, head and neck in the week prior to Treatment Days 1 through Day 6 of the Treatment Period
* Has illness or history of illness which might confound study results or pose unwarranted risk
* Known history of QT interval prolongation
* Uses illicit drugs or abuses alcohol
* Mentally incapacitated or has a significant emotional or psychiatric disorder
* History of hypersensitivity to aprepitant, ondansetron or dexamethasone
* Pregnant or breast-feeding
* Has participated in a study with aprepitant or taken a non-approved (investigational) drug within the last 4 weeks
* Has concurrent condition, such as systemic fungal infection or uncontrolled diabetes, that precludes administration of dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2012-09-24 (Actual); Primary Completion 2014-11-03 (Actual); Study Completion 2014-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Weinstein C, Jordan K, Green SA, Camacho E, Khanani S, Beckford-Brathwaite E, Vallejos W, Liang LW, Noga SJ, Rapoport BL. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with moderately emetogenic chemotherapy: results of a randomized, double-blind phase III trial. Ann Oncol. 2016 Jan;27(1):172-8. doi: 10.1093/annonc/mdv482. Epub 2015 Oct 8. PMID 26449391
- [Derived] Weinstein C, Jordan K, Green S, Khanani S, Beckford-Brathwaite E, Vallejos W, Pong A, Noga SJ, Rapoport BL. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting in patients receiving moderately emetogenic chemotherapy regimens: a subgroup analysis from a randomized clinical trial of response in subjects by cancer type. BMC Cancer. 2020 Sep 25;20(1):918. doi: 10.1186/s12885-020-07259-5. PMID 32988373
- [Derived] Weinstein C, Jordan K, Green SA, Camacho E, Khanani S, Beckford-Brathwaite E, Pong A, Noga SJ, Rapoport BL. Evaluation of factors contributing to the response to fosaprepitant in a heterogeneous, moderately emetogenic chemotherapy population: an exploratory analysis of a randomized phase III trial. Support Care Cancer. 2018 Nov;26(11):3773-3780. doi: 10.1007/s00520-018-4242-x. Epub 2018 May 28. PMID 29808377
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0517-031&kw=0517-031&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14 participants did not receive any study drug: 4 in the Fosaprepitant Regimen and 10 in the Control Regimen. One participant who was randomized to the Control Regimen received the Fosaprepitant Regimen.
Groups:
- Fosaprepitant Regimen: On Day 1, participants received fosaprepitant, 150 mg intravenous (IV) infusion, ~30 minutes prior to chemotherapy PLUS dexamethasone 12 mg, orally (PO) ~30 minutes prior to chemotherapy PLUS ondansetron 16 mg total dose: 8 mg PO ~30-60 minutes prior to chemotherapy, followed by 8 mg PO, 8 hours after first dose PLUS dexamethasone placebo, PO ~30 minutes prior to chemotherapy. On Days 2 and 3, participants received ondansetron placebo, PO every 12 hours. Rescue Therapy: For established cases of nausea or vomiting, medications may have been prescribed from these permitted choices: 5-hydroxytryptamine 3 (5-HT3) antagonists (granisetron, dolasetron, tropisetron or ondansetron); phenothiazines (e.g. prochlorperazine, fluphenazine, perphenazine, thiethylperazine, or chlorpromazine); butyrophenones (e.g. haloperidol or droperidol); benzamides (e.g. metoclopramide or alizapride); benzodiazepines; corticosteroids; domperidone.
Period: Overall Study
Arm/Group | Fosaprepitant Regimen | Control Regimen
Started | 507 | 508
Treated | 503 | 498
Completed | 485 | 490
Not Completed | 22 | 18
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Non-compliance with Protocol | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 9 | 3
Not completed — Not Treated | 4 | 10
Not completed — Lost Source Documentation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline analysis population is consistent with the Intent-to-Treat (ITT) population, i.e., all randomized participants who received ≥1 dose of study drug within the assigned treatment regimen. Note: One participant with missing source documentation in the Fosaprepitant Regimen was excluded from the ITT population.
Groups:
- Fosaprepitant Regimen: On Day 1, participants received fosaprepitant, 150 mg IV infusion, ~30 minutes prior to chemotherapy PLUS dexamethasone 12 mg, PO ~30 minutes prior to chemotherapy PLUS ondansetron 16 mg total dose: 8 mg PO ~30-60 minutes prior to chemotherapy, followed by 8 mg PO, 8 hours after first dose PLUS dexamethasone placebo, PO ~30 minutes prior to chemotherapy. On Days 2 and 3, participants received ondansetron placebo, PO every 12 hours. Rescue Therapy: For established cases of nausea or vomiting, medications may have been prescribed from these permitted choices: 5-HT3 antagonists (granisetron, dolasetron, tropisetron or ondansetron); phenothiazines (e.g. prochlorperazine, fluphenazine, perphenazine, thiethylperazine, or chlorpromazine); butyrophenones (e.g. haloperidol or droperidol); benzamides (e.g. metoclopramide or alizapride); benzodiazepines; corticosteroids; domperidone.
- Total: Total of all reporting groups
Arm/Group | Fosaprepitant Regimen | Control Regimen | Total
Number analyzed (Participants) | 502 | 498 | 1000
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (11.8) | 59.1 (12.3) | 59.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 293 | 591
  Male | 204 | 205 | 409

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response From 25 to 120 Hours After Initiation of Moderately Emetogenic Chemotherapy (MEC)
Description: A Complete Response was defined as no vomiting and no use of rescue medication.
Time Frame: 25 to 120 hours after initiation of MEC
Population: The ITT population consisted of all randomized participants who received ≥1 dose of study drug within the assigned treatment regimen. One participant in the Fosaprepitant Regimen was excluded from the ITT population due to missing source documentation. One participant in the Control Regimen was treated with fosaprepitant in error.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen | Control Regimen
Number analyzed (Participants) | 502 | 498
Percentage of Participants | 78.9 | 68.5
Statistical Analysis 1: Comparison: Fosaprepitant Regimen vs Control Regimen; Percentage difference in Fosaprepitant Regimen vs. Control Regimen; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value based on Cochran-Mantel-Haenszel (CMH) method with stratification of gender

2. Primary Outcome: Percentage of Participants With Infusion-site Thrombophlebitis
Description: The percentages of participants with infusion-site thrombophlebitis are presented. Thrombophlebitis was defined as a condition affecting a superficial vein used for an IV infusion, associated with red color, hardness upon palpation, and the presence of a tender cord and possible fever.
Time Frame: Day 1 through Day 17, inclusive
Population: The Safety population consisted of all randomized participants who received study drug as treated.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen | Control Regimen
Number analyzed (Participants) | 504 | 497
Percentage of Participants | 0.6 | 0.0
Statistical Analysis 1: Comparison: Fosaprepitant Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.085, Miettinen & Nurminen method — P-value based on Miettinen & Nurminen method; Difference in percentage vs. Control = 0.6, 95% CI 2-sided [-0.2 to 1.7]

3. Primary Outcome: Percentage of Participants With Severe Infusion-site Reactions
Description: The percentages of participants with severe infusion-site reactions, including severe site pain, or severe site redness (erythema) or severe site hardness (induration) are presented.
Time Frame: Day 1 through Day 17, inclusive
Population: The Safety population consisted of all randomized participants who received study drug as treated.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen | Control Regimen
Number analyzed (Participants) | 504 | 497
Percentage of Participants | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants With Complete Response From 0 to 120 Hours After Initiation of MEC
Description: A Complete Response was defined as no vomiting and no use of rescue medication.
Time Frame: 0 to 120 hours after initiation of MEC
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen | Control Regimen
Number analyzed (Participants) | 502 | 498
Percentage of Participants | 77.1 | 66.9
Statistical Analysis 1: Comparison: Fosaprepitant Regimen vs Control Regimen; Percentage difference in Fosaprepitant Regimen vs. Control Regimen; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value based on CMH method with stratification of gender

5. Secondary Outcome: Percentage of Participants With Complete Response From 0 to 24 Hours After Initiation of MEC
Description: A Complete Response was defined as no vomiting and no use of rescue medication.
Time Frame: 0 to 24 hours after initiation of MEC
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen | Control Regimen
Number analyzed (Participants) | 502 | 498
Percentage of Participants | 93.2 | 91.0
Statistical Analysis 1: Comparison: Fosaprepitant Regimen vs Control Regimen; Percentage difference in Fosaprepitant Regimen vs. Control Regimen; Test type: Superiority or Other; p = 0.184, Cochran-Mantel-Haenszel — P-value based on CMH method with stratification of gender

6. Secondary Outcome: Percentage of Participants With No Vomiting From 0 to 120 Hours After Initiation of MEC
Description: No Vomiting was defined as no emetic (vomiting) episodes, including no vomiting and no retching or dry heaves (attempts to vomit that are not productive of stomach contents), regardless of use of rescue medication.
Time Frame: 0 to 120 hours after initiation of MEC
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Fosaprepitant Regimen | Control Regimen
Number analyzed (Participants) | 502 | 498
Percentage of participants | 82.7 | 72.9
Statistical Analysis 1: Comparison: Fosaprepitant Regimen vs Control Regimen; Percentage difference in Fosaprepitant Regimen vs. Control Regimen; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value based on CMH method with stratification of gender

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 17, inclusive (Up to 2 weeks after last dose of study drug)
Description: The Safety population consisted of all participants who received study drug. Participants are included in the treatment group based on the study drug they actually received.
Arm/Group | Fosaprepitant Regimen | Control Regimen
Serious Adverse Events (participants affected / at risk) | 39/504 | 35/497
Other Adverse Events (participants affected / at risk) | 190/504 | 193/497
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant Regimen (N=504) | Control Regimen (N=497)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant Regimen (N=504) | Control Regimen (N=497)
Neutropenia (Blood and lymphatic system disorders) | 38 (38) | 33 (33)
Constipation (Gastrointestinal disorders) | 47 (48) | 51 (53)
Diarrhoea (Gastrointestinal disorders) | 63 (66) | 55 (57)
Fatigue (General disorders) | 75 (78) | 64 (64)
Decreased appetite (Metabolism and nutrition disorders) | 26 (27) | 32 (32)
Headache (Nervous system disorders) | 30 (32) | 35 (37)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.